CLINICAL TRIAL: NCT03630198
Title: The Use of Local Anesthetic in Intralesional Corticosteroid Injections; A Randomized, Double Blind Controlled Trial
Brief Title: Pain Outcomes Following Intralesional Corticosteroid Injections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Brian Drolet, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 181119
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Results first posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-02

CONDITIONS: Keloid; Alopecia Areata; Acne; Hypertrophic Scar; Epidermal Inclusion Cyst; Frontal Fibrosing Alopecia; Lichen Plano-Pilaris; Keratoacanthoma; Plaque Psoriasis; Lichen Simplex Chronicus; Prurigo Nodularis; Nummular Eczema; Granuloma Annulare; Morphea; Lichen Planus
Keywords: corticosteroid; local anesthetic
MeSH Terms: conditions — Keloid; Alopecia Areata; Acne Vulgaris; Cicatrix, Hypertrophic; Dermoid Cyst; Lichen Planus; Keratoacanthoma; Neurodermatitis; Granuloma Annulare; Scleroderma, Localized | interventions — Adrenal Cortex Hormones; Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Corticosteroid with lidocaine (Active Comparator): This arm will include an injection mixture of corticosteroid and lidocaine
  Interventions: Drug: Corticosteroid with lidocaine
- Corticosteroid with normal saline (Experimental): This arm will include a mixture of corticosteroid and normal saline. The purpose of normal saline is to keep the volume and concentration similar when compared to the injections containing lidocaine.
  Interventions: Drug: Corticosteroid with normal saline

INTERVENTIONS:
Drug: Corticosteroid with lidocaine — Intralesional corticosteroid injection
  Arms: Corticosteroid with lidocaine
Drug: Corticosteroid with normal saline — Intralesional corticosteroid injection
  Arms: Corticosteroid with normal saline

SUMMARY:
Corticosteroid therapy, including intralesional and topical applications, has many indications within the fields of Dermatology, Plastic Surgery, and Orthopedics. However, these injections can be quite painful, which leads many patients to discontinue treatment.

Often, the injection involves a mixture of local anesthetic and corticosteroids despite a lack of evidence that the use of lidocaine improves pain. Due to the acidic pH, the lidocaine component of the injection can actually cause a significant burning sensation during the procedure. Lidocaine does not have anti-inflammatory properties and does not treat the underlying pathology. By including another medication, lidocaine also adds cost and risk to the procedure.

The purpose of this study is to see if removing lidocaine from intralesional injections decreases the pain of injection.

ELIGIBILITY:
Inclusion Criteria:

* >12 years old presenting with an indication for intralesional steroid injection

Exclusion Criteria:

* Unconsentable
* Not a candidate for corticosteroid injection
* Contraindication to lidocaine

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Drolet, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers

REFERENCES:
- [Derived] Zakria D, Patrinely JR Jr, Dewan AK, Albers SE, Wheless LE, Simmons AN, Drolet BC. Intralesional corticosteroid injections are less painful without local anesthetic: a double-blind, randomized controlled trial. J Dermatolog Treat. 2022 Jun;33(4):2034-2037. doi: 10.1080/09546634.2021.1906842. Epub 2021 Apr 7. PMID 33760691

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Corticosteroid With Lidocaine | Corticosteroid With Normal Saline
Started | 13 | 18
Completed | 13 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Corticosteroid With Lidocaine | Corticosteroid With Normal Saline | Total
Number analyzed (Participants) | 13 | 18 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 18 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (18.2) | 52 (19.2) | 43 (20.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 7 | 8 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 18 | 31

OUTCOME MEASURES:

1. Primary Outcome: Pain Outcome: Visual Analog Scale
Description: Assessed using the visual analog scale (0-10 scale). Zero indicates no pain, 10 indicates worst pain ever.
Time Frame: Assessed 1 minute after the injection (in clinic)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Corticosteroid With Lidocaine | Corticosteroid With Normal Saline
Number analyzed (Participants) | 13 | 18
Score on a scale | 5.4 (2.4) | 2.7 (2.3)

2. Post Hoc Outcome: Pain Outcome: Visual Analog Scale
Description: Assessed using the visual analog scale (0-10 scale). Zero indicates no pain, 10 indicates worst pain ever.
Time Frame: Assessed at 6 hours and 24 hours after injection
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Corticosteroid With Lidocaine | Corticosteroid With Normal Saline
Number analyzed (Participants) | 13 | 18
Score on a scale
  Pain (6 hour) | 0.9 (2.1) | 0.1 (1.5)
  Pain (24 hour) | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 1 year after injection
Description: No difference
Arm/Group | Corticosteroid With Lidocaine | Corticosteroid With Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/18
Other Adverse Events (participants affected / at risk) | 0/13 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT03630198/Prot_SAP_000.pdf